CLINICAL TRIAL: NCT00238381
Title: Clinical Function After Total Mesorectal Excision and Rectal Replacement. A Prospective Randomized Trial Comparing Side-to-End Anastomosis, Colon-J-Pouch and Straight Coloanal Anastomosis
Brief Title: Rectal Reconstruction in Treating Patients Who Are Undergoing Surgery for Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 40/04; EU-20528
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage 0 rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Other): Patients undergo total mesorectal excision (TME) by standard methods or laparoscopically and side-to-end anastomosis rectal reconstruction.
  Interventions: Procedure: side-to-end anastomosis
- Arm II (Other): Patients undergo TME and colon-J-pouch anastomosis rectal reconstruction.
  Interventions: Procedure: 5 cm colon-J-pouch
- Arm III (Other): Patients undergo straight coloanal anastomosis with/without temporary protective ileostomy
  Interventions: Procedure: straight coloanal anastomosis

INTERVENTIONS:
Procedure: 5 cm colon-J-pouch — 5 cm colon-J-pouch with/without temporary protective ileostomy
  Arms: Arm II
Procedure: side-to-end anastomosis — side-to-end anastomosis with/without temporary protective ileostomy
  Arms: Arm I
Procedure: straight coloanal anastomosis — straight coloanal anastomosis with/without temporary protective ileostomy
  Arms: Arm III

SUMMARY:
RATIONALE: Rectal reconstruction after surgery to treat rectal cancer may help patients keep some of their bowel function. It is not yet known which method of rectal reconstruction is most effective after surgery.

PURPOSE: This randomized phase III trial is studying three different methods of rectal reconstruction to compare how well they work in treating patients who are undergoing surgery for rectal cancer.

DETAILED DESCRIPTION:
This is a randomized, multicenter study. Patients are stratified according to participating center, gender, distance of the distal tumor margin from the dentate line (> 5 cm vs ≤ 5 cm), age (< 70 vs ≥ 70), neoadjuvant chemoradiotherapy (yes vs no), and distant metastasis (M0 vs M1). Patients are randomized to 1 of 3 treatment arms.

ELIGIBILITY:
* Histologically proven rectal adenocarcinoma or rectal adenoma with/without neoadjuvant radiochemotherapy
* Total mesorectal excision needed
* Age ≥ 18 years
* Clinically normal function of the sphincter muscles (no history of frequent fecal incontinence for liquid or solid stools)
* Any T, any N, any M or adenoma
* An R0-resection is expected (liver metastases planned to be simultaneously
* Written informed consent, signed and dated by the patient and the investigator
* Completed baseline quality of life questionnaire

Exclusion criteria:

* Rectal tumor other than adenocarcinoma or adenoma
* Previous rectal cancer surgery, other than local excision within the last 2 months
* Histologically proven chronic inflammatory bowel disease
* Contraindications to any of the 3 surgical techniques
* BMI > 35
* Patients with psychiatric, addictive or any disorder that would prohibit the understanding and giving of informed consent, completing the QL questionnaires and/or following the structured interview
* Inability to read and understand any of the languages available on the QL questionnaires,and spoken during the interview (German, French, Italian)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2005-07; Primary Completion 2014-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Composite evacuation score after total mesorectal excision | 12 months after surgery

SECONDARY OUTCOMES:
Composite evacuation score at 6, 18, and 24 months after total mesorectal excision | 6, 18 and 24 months after surgery
Composite incontinence score after total mesorectal excision | 6, 12, 18 and 24 months
Quality of life after total mesorectal excision | 6, 12m 18 and 24 months
Overall survival | 2 years follow-up
Morbidity | 2 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christian T. Hamel, MD, Study Chair — Kantonsspital - Abteilung Onkologie; Walter R. Marti, Prof., Study Chair — Kantonsspital Aarau; Markus Zuber, MD, Study Chair — Kantonsspital Olten
Locations (18):
- Kreiskrankenhaus Lörrach, Loerrach, Germany
- Switzerland (17):
  - Kantonsspital Aarau, Aarau
  - Zuger Kantonsspital AG, Baar
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Bezirksspital Dornach, Dornach
  - Hopitaux Universitaires de Geneve, Geneva
  - Hopital de La Chaux-de-Fonds, La Chaux-de-Fonds
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Luzerne
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital Olten, Olten
  - GZO Spital Wetzikon, Wetzikon
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Marti WR, Curti G, Wehrli H, Grieder F, Graf M, Gloor B, Zuber M, Demartines N, Fasolini F, Lerf B, Kettelhack C, Andrieu C, Bigler M, Hayoz S, Ribi K, Hamel C; Swiss Group for Clinical Cancer Research (SAKK), Section Surgery. Clinical Outcome After Rectal Replacement With Side-to-End, Colon-J-Pouch, or Straight Colorectal Anastomosis Following Total Mesorectal Excision: A Swiss Prospective, Randomized, Multicenter Trial (SAKK 40/04). Ann Surg. 2019 May;269(5):827-835. doi: 10.1097/SLA.0000000000003057. PMID 30252681